CLINICAL TRIAL: NCT03065595
Title: The Effect of Ophicephalus Striatus Extract on Levels of Insulin-like Growth Factor-1 (IGF-1), Albumin, and Mini Nutritional Assessment Score in Elderly Patients With Malnutrition: A Double Blind Randomized Controlled Trial
Brief Title: The Effect of Ophiocephalus Striatus Extract on Levels of IGF-1, Albumin, and MNA Score in Elderly With Malnutrition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Roza Mulyana, MD, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16268
Record Dates: First submitted 2017-02-19; First posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Malnutrition
Keywords: Ophiocephalus striatus; IGF-1; hypoalbuminemia; MNA score; elderly
MeSH Terms: conditions — Malnutrition; Hypoalbuminemia

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Placebo Comparator): Ophicephalus striatus extract
  Interventions: Dietary Supplement: Ophiochepalus striatus extract
- Control (Active Comparator): Placebo drug
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ophiochepalus striatus extract — each sachet of ophiochepalus striatus extract is poured into 50 mL normal water and drink two times/day
  Other Names: VIP ALBUMIN
  Arms: Intervention
Other: Placebo — each sachet of placebo drug is poured into 50 mL normal water and drink two times/day
  Arms: Control

SUMMARY:
This study is a double-blind randomized controlled trial comparing the effect of Ophiocephalus striatus extract in elderly patients with malnutrition. The measured outcomes are the level of IGF-1, albumin, and MNA score.

DETAILED DESCRIPTION:
This research was conducted in Cipto Mangunkusumo General Hospital and M. Djamil General Hospital, in collaboration with Biomedical Laboratory Faculty of Medicine University of Andalas and Prodia Laboratory, Indonesia. The inclusion criteria were elderly patients (≥ 60 y.o.) with malnutrition (MNA score ≤ 23,5) and hypoalbuminaemia (< 3,5 g/dL), had been treated, and permitted to leave from the hospital. All participants had been interviewed and physically examined to measure the anthropometric profile. Investigators also measured participant's Activity of Daily Living ADL Barthel, Geriatric Depression Scale (GDS), and Abbreviated Mental Test (AMT) to assess participant's compliance for consuming Ophiocephalus striatus extract. Blood samples were obtained to measure participant's level of IGF-1 and albumin before intervention.

Recruited-randomized participants were classified into two groups (control and intervention) with double-blind scheme. Intervention group was given the extract 5 grams two times/day for two weeks. After two weeks, all participants were invited back to out-patient clinic in hospital. MNA score was measured after the intervention. Blood sample were obtained again to know if there were any changes in IGF-1 level and albumin level.

Finally, investigators analyzed results to generate the conclusion.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patient (≥ 60 y.o.)
* Malnutrition or high risk for malnutrition (MNA score ≤ 23,5)
* Hypoalbunemia (albumin level < 3,5 g/dL)

Exclusion Criteria:

* chronic liver disease (liver cirrhosis) or severe liver dysfunction or increasing ALT > 3x normal
* renal dysfunction with glomerulus filtration rate (< 30mL/minute)
* nephrotic syndrome
* acute infection / stroke / trauma
* neoplasma
* depression with Geriatric Depression Scale > 10
* hypersensitivity to Ophiocephalus striatus
* receive parenteral albumin
* refuse to accept the treatment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-02-14 (Actual)

PRIMARY OUTCOMES:
Serum IGF-1 | 2 weeks
  IGF-1 will be measured from blood serum. The level will be compared between intervention and control group (ng/mL)
Serum albumin | 2 weeks
  Albumin will be measured from blood serum. The level will be compared between intervention and control group (g/dL)
MNA score | 2 weeks
  MNA score was measured from direct anamnesis to the patient (or family) and anthropometric profile.

IPD SHARING:
Plan to Share IPD: Yes
The research findings will be disseminated via publication of results, submission of information to public accessible databases, or meetings